CLINICAL TRIAL: NCT03014466
Title: Screen-Based Distraction Tool for Preoperative Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-37577
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet (Active Comparator): Preoperative patients will utilize a video tablet for addressing pre anesthesia anxiety
  Interventions: Behavioral: Use of Video Tablet
- Video Projector (Experimental): Preoperative patients will utilize a video projection unit for addressing pre anesthesia anxiety
  Interventions: Behavioral: Use of Video Projector

INTERVENTIONS:
Behavioral: Use of Video Projector — Bed mounted video projector that is used to play videos of the patient's choosing prior to induction of anesthesia
  Other Names: Bedside Entertainment Theater
  Arms: Video Projector
Behavioral: Use of Video Tablet — 7 inch video tablet that is used for displaying videos of the patient's choosing prior to induction of anesthesia
  Arms: Tablet

SUMMARY:
Preoperative anxiety in pediatric patients undergoing surgical procedures has been previously shown to increase the likelihood of family stressors, post- operative pain, agitation, sleep disturbances, and negative behavioral changes. The purpose of this study is to determine whether the use of a bed mounted Video Projection unit (i.e. BERT, Bedside EnterRtainment Theater) is more effective than the use of a standard of care tablet (i.e., iPad) for preventing anxiety before surgery among children undergoing anesthesia and surgery. The anticipated primary outcome will be reduction of child's anxiety in the preoperative and operating room setting and compliance with mask induction.

DETAILED DESCRIPTION:
Patients will initially be approached about the study during a pre-surgical phone call that every patient receives prior to their procedure by a Nurse Practitioner (NP). During this phone call, the NP will ask if the family would be interested in participating in a research study and if they may be contacted by the research team. If the family expresses interest, the NP will follow-up with the research team and a eligibility screening phone call will be given. If families decline interest, we will respect their decision and will not pursue the family any further for this study. Not all families will be available during the initial pre- surgical phone call, and in this case, the medical staff member and research assistant will approach the family in the pre-operative holding area day of surgery. Interested families will be given a brochure with information about the study and screened for eligibility.

Upon arrival for preoperative preparations, the research assistant will go over the consent and assent forms with the parent and child and answer any questions they may have about the study. While child is being prepped to be transported to the preoperative holding area, a research staff member will determine whether the participant will receive the standard care (i.e. entertainment via tablet) or the (i.e. BERT, Bedside EnteRtainment System; Video Projection) via random assignment. Once determined, the research staff will set up the system for the patient and will be asked to fill out questionnaires, on REDCap or by paper, about how they are feeling at that time before their surgery. Parents will also be asked to fill out questionnaires about their feelings of their child's preoperative emotions. The child will continue to view their preoperative entertainment through to induction. A video camera mounted to the BERT screen or tablet will be used for retrospective coding by blinded research assistants. When possible, a blinded research assistant will also live-code the observer-rated surveys. We aim for this to occur for around 20-30% of participants. care) The research assistants will complete the mYPAS (modified Yale Preoperative Anxiety Scale) and ICC (Induction Compliance Checklist) when coding in vivo. Vitals (i.e. blood pressure, heart rate, oxygen saturation, end tidal CO2, and temperature) will also be recorded as they undergo preoperative preparations. The parent will be asked to remain with their child from the preoperative holding area until the child has undergone induction. Once child enters induction phase in the OR, the patient will undergo surgery as scheduled.

Post-operation, the research assistant will further examine the child's behaviors as they wake from anesthesia. They will also give the the parent, child, and child's anesthesiologist a survey about their experiences with the screen-based device. 1 week after the surgery, the research assistant will follow up with the parent/guardian with questions about their and their child's preoperative and perioperative via phone. The call will also be audio recorded. After the one-week follow-up survey, the study will be concluded for the participant.

b) Explain how the above research procedures are the least risky that can be performed consistent with sound research design.

All survey questions are meant to answer questions pertaining to the study aims. Set up of the Video Projection unit will be performed by trained members of the research team and will be of minimal risk to patients.

The risks associated with this study include the possibility of participation being discovered by others outside of the study team. This is highly unlikely given the precautions that will be described later in this application.

c) State if deception will be used. If so, provide the rationale and describe debriefing procedures. Since you will not be fully informing the participant in your consent process and form, complete an alteration of consent (in section 13). Submit a debriefing script (in section 16).

Deception will not be used.

d) State if audio or video recording will occur. Describe what will become of the recording after use, e.g., shown at scientific meetings, erased. Describe the final disposition of the recordings.

Participants will be video taped to capture the patient's full experience with the Video Projection unit and its effect during preoperative and perioperative procedure. The video camera will be mounted on the tablet or BERT system. Videos will be coded by the research team, and will not contain PHI. Audio will be recorded from the follow-up phone calls so that the parents' responses will be fully captured in our measures. These videos and audio files will be stored on a secured, password protected, and encrypted computer, which only authorized members of the study will have access to. The videos and audio files will be destroyed 6 years after the publication of the study. These videos and audio files may be presented at scientific meetings and this will be included in the consent.

e) Describe alternative procedures or courses of treatment, if any, that might be advantageous to the participant. Describe potential risks and benefits associated with these. Any standard treatment that is being withheld must be disclosed in the consent process and form. (i.e. standard-of-care drug, different interventional procedure, no procedure or treatment, palliative care, other research studies).

This is a randomized trial to validate the effectiveness of using a Video Projection unit, therefore there will be subjects that undergo standard treatment as a result of the randomization. The randomization will be performed by the research assistant following consent. Parents must be with their child from the pre-operative area until induction. They will have the option to opt-out of the study if the parent or child does not want the parent present or there is a strong patient or parent preference for pharmacological anxiolytic or a specific anxiety-reduction technique.

f) Will it be possible to continue the more (most) appropriate therapy for the participant(s) after the conclusion of the study?

N/A. The interventional technologies will only be implemented to allay preoperative anxiety, therefore will not be continued after the surgery.

g) Study Endpoint. What are the guidelines or end points by which you can evaluate the different treatments (i.e. study drug, device, procedure) during the study? If one proves to be clearly more effective than another (or others) during the course of a study, will the study be terminated before the projected total participant population has been enrolled? When will the study end if no important differences are detected?

The endpoint of the study will be determined by the completion of the target number of participants. The target number of participants for the study is 30 participants in each randomized group (i.e. standard care tablet and Video Projection unit group) for a total of 60 patients who complete the study.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. be between ages of 4-10 years of age
2. have comprehension of instructions in the English language
3. have parental consent
4. Pediatric patient must be undergoing non-emergent outpatient surgery at Lucile Packard Children's Hospital
5. Children who are normally healthy (ASA I) or have a mild systemic disease (ASA II) -

Exclusion Criteria:

General Exclusion Criteria are as follows:

1. Significant cognitive impairment/developmental delays per parental report or H&P.
2. Children with ASA III, ASA IV (severe systemic disease that is a constant threat to life) or ASA V (unstable patients not expected to survive >24hours or without the operation)
3. Children currently taking psychotropic mediations will be excluded from this study due to the affect emotion modulation
4. Strong parental or patient preference for pharmacological anxiolytic
5. Strong parental or patient preference for specific anxiety-reducing technique
6. Children born before 32 week gestation
7. Any indication that the patient may be admitted post-operatively
8. Child has had previous surgery or has undergone general anesthesia
9. Parent does not want to be present during transport to the OR or during induction -

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Anxiety at Induction of Anesthesia | 30 minutes
  Modified Yale Perioperative Anxiety Score at induction of anesthesia. This is a validated scale used to assess patient periprocedural anxiety

SECONDARY OUTCOMES:
Induction Compliance | 5 minutes
  Validated score for assessing patient compliance with anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Rodriguez, MD, Principal Investigator — Stanford School of Medicine

IPD SHARING:
Plan to Share IPD: No